CLINICAL TRIAL: NCT00368186
Title: An Open, Multicenter Clinical Trial to Investigate the Immunogenicity and Safety of the Pneumococcal 7-Valent Conjugate Vaccine (PREVENAR) in Sickle Cell Disease Infants.
Brief Title: Immunogenicity and Safety Study of Pneumococcal 7-Valent Conjugate Vaccine in Sickle Cell Disease Infants.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0877X-100722
Record Dates: First submitted 2006-08-21; First posted 2006-08-24 (Estimated); Last update posted 2006-08-24 (Estimated); Status verified 2006-08

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

INTERVENTIONS:
Biological: Pneumo 23

SUMMARY:
The primary objectives of this study were to assess the immunogenicity and the tolerance of the heptavalent pneumococcal conjugate vaccine (Prevenar) in young infants (2 months of age) with sickle cell disease when administred at 2,3, and 4 months of age.

ELIGIBILITY:
Inclusion Criteria

Infants with neonatal diagnosis of sickle cell disease and confirmed hemoglobin status by hemoglobin electrophoresis.

Exclusion Criteria

Previous immunization with pneumococcal-containing vaccines.

History of pneumococcal invasive disease (meningitis, bacteremia, pneumonia).

Known or suspected impairments of the immune system (including HIV infection) or recipients of immuno-suppressant agents.

Other Exclusions apply.

Ages: 57 Days to 112 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51
Dates: Start 2001-05; Study Completion 2002-11

PRIMARY OUTCOMES:
Antibody responses to pneumococcal capsular polysaccharides antigens contained in PCV7 vaccine; local and systemic reactions.

SECONDARY OUTCOMES:
Opsonophagocytic activity; S. pneumoniae nasopharyngeal carriage.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Paris, France